CLINICAL TRIAL: NCT01076036
Title: CorPath™ 200 System: Coronary Remote Catheterization Feasibility Study
Brief Title: CorPath™ 200: Robotically-Assisted Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Corindus-Corbic-2010
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease
Keywords: ischemia; stent
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CorPath 200 System (Experimental): Robotic-assisted PCI with the CorPath 200
  Interventions: Device: CorPath 200

INTERVENTIONS:
Device: CorPath 200 — CorPath™ 200 robotically-assisted percutaneous coronary intervention
Device: CorPath 200 — CorPath PCI - robotic-assisted percutaneous coronary intervention

SUMMARY:
An open-label, prospective, single-arm study is designed to evaluate safety, clinical and technical efficacy of the CorPath 200 System in delivery and manipulation of the coronary guide wires and balloon/stent systems for use in robotically-assisted, percutaneous coronary intervention (PCI) procedures.

DETAILED DESCRIPTION:
Objective The study objective was to evaluate the safety and technical efficacy of the CorPath 200 System in delivery and manipulation of commercially available coronary guidewires and rapid exchange balloon/stent catheter for use in percutaneous coronary interventions (PCI).

I. Primary Endpoints A. Efficacy Device Clinical Success: Achievement of a < 30% final diameter stenosis after utilizing the CorPathTM 200 System to deliver a PTCA balloon and then stent to the target lesion, and successfully retract the devices without the occurrence of any In-Hospital MACE (Major Adverse Cardiac Event) evaluated at 48 hours post procedure or hospital discharge, whichever occurs first.

B. Safety In-Hospital MACE: Defined as the composite of death (all cause mortality), recurrent MI, and target vessel revascularization (emergent coronary artery bypass surgery [CABG] or PCI) evaluated at 48 hours post procedure or hospital discharge, whichever occurs first.

II. Secondary Endpoints A. Efficacy CorPath Success: Ability to navigate the guide wire and balloon/stent system utilizing the CorPath™ device to the target site without the occurrence of any In-Hospital MACE, evaluated at 48 hours post index procedure or hospital discharge, whichever occurs first.

Subject Clinical Success: Achievement of a <30% final diameter stenosis of target lesion after treatment with PTCA/coronary stent without the occurrence of any In-Hospital MACE, evaluated at 48 hours post-index procedure or hospital discharge, whichever occurs first.

B. Safety:

MACE at 30 Days: Defined as the composite of death, recurrent MI and/or target vessel revascularization (emergent coronary artery bypass surgery [CABG] or PCI) evaluated at 30 days post index procedure.

Adverse Events:

A summary of all adverse events observed in the trial summarized as either serious or non-serious and summarized by attribution.

C. Clinical Utility

Procedure Attributes:

* Reduction in radiation exposure to the primary operator based on radiation dosimetry measurements at the procedure table and on a primary operator.
* Total Procedure time based on the time of insertion of hemostasis sheath through the time of final guide catheter withdrawal.

CorPath Device Attributes:

Subjective assessment by the operator of the following device performance attributes:

* Movement of the guide wire (rotating and advancing) to the target.
* Maneuvering and position of the guide wire to the target.
* Movement of the stent/balloon (advancing) to the target.
* Ability to deliver the PTCA/stent system to the intended target lesion.
* Ease of use of the system by the interventional team.

Material & Methods Corindus obtained approval (from the CORBIC Ethics Committee and INVIMA - Colombian Ministry of Health) in 2009 to conduct the clinical study "CorPath™ 200 System: Coronary Remote Catheterization Feasibility Study" at CORBIC Cardio-Neuro-Vascular Institute, Envigado, Colombia.

The study is a single arm, open label, prospective registry to treat a de novo lesion (2.5 mm - 4.0 mm in diameter, 25.0 mm in length with >50% stenosis) utilizing the CorPath 200 System to deliver, manipulate and retrieve a guidewire and a balloon/stent catheter system.

ELIGIBILITY:
General Inclusion Criteria:

* The subject is an acceptable candidate for PCI.
* The subject must have clinical evidence of ischemic heart disease or a positive functional study.
* Female subjects must be of non-child bearing potential, or if able to bear children, have a negative pregnancy test within seven (7) days prior to index procedure.
* The subject or the legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent.

Angiographic Inclusion Criteria:

* Study lesion is de novo native coronary artery lesion (i.e., a coronary lesion not previously treated)
* The study lesion is intended to be treated with one stent. Maximum stent length allowed is 20 mm.
* The study reference vessel diameter is between 2.50 mm and 4.5 mm by visual estimate.
* Study lesion diameter showing significant stenosis of at least 50% by visual estimate.

General Exclusion Criteria:

* Subject requires planned PCI or CABG within 30 days following the index procedure.
* Subject has evolving ST elevation myocardial infarction (STEMI) (i.e., beginning of MI symptoms within 72 hours prior to the planned index procedure).
* Subject has documented left ventricular ejection fraction < 30%.
* Subject has known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, stainless steel, or a sensitivity to contrast media, which cannot be adequately pre-medicated.
* Subject has a platelet count < 100,000 cell/mm3 or > 700,000 cell/ mm3, a WBC of < 3000 cell/ mm3 (e.g. thrombocytopenia, thrombocythemia, neutropenia or leucopenia).
* Subject has a history of a stroke (CVA) or TIA within 30-days prior to planned index procedure.
* Subject has an active peptic ulcer or upper GI bleeding within the 6 months prior to planned index procedure.
* Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Subject is currently participating in another investigational drug l drug or device trial that has not completed the entire follow up period.

Angiographic Exclusion Criteria:

* Study lesion that cannot be fully covered by a single stent of maximal length
* Subject requires treatment of multiple lesions in the study vessel at the time of index procedure.
* The study lesion requires planned treatment with DCA, laser, rotational atherectomy, or any device except for balloon dilatation prior to stent placement.
* The study vessel has evidence of intraluminal thrombus or moderate to severe tortuosity (> 90o) proximal to the target lesion.
* The study lesion has any of the following characteristics:

  1. Total occlusion
  2. Ostial location
  3. Involves a side branch > 2.0 mm vessel diameter
  4. Is located at >45° bend in the vessel
  5. Is moderately to severely calcified
  6. Moderate-to-severe calcification at the part of the vessel prior to target lesion
* Unprotected left main coronary artery disease (an obstruction greater than 50% diameter stenosis in the left main coronary artery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Granada, MD, Principal Investigator — CORBIC and CRF
Locations (1):
- CORBIC Cardio-Neuro-Vascular Institute, Medellín, Colombia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February-March 2011 at CORBIC, Envigado, Colombia
Groups:
- Group 1: Group 1 was treated using the CorPath device.
Period: Overall Study
Arm/Group | Group 1
Started | 10
# of Procedures | 8
Complete CorPath Procedures | 8
Completed | 8
Not Completed | 2
Not completed — Didn't meet inclusion/exclusion criteria | 2

BASELINE CHARACTERISTICS:
Groups:
- Investigational: CorPath® 200 System
Arm/Group | Investigational
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  Colombia | 8

OUTCOME MEASURES:

1. Primary Outcome: Clinical Procedural Success
Description: The percentage of Participants with <30% final diameter stenosis of the target lesion without in-hospital major adverse cardiovascular events (MACE) (defined as the composite of death, recurrent MI, and target vessel revascularization)
Time Frame: 48-hrs or hospital discharge, whichever occurs first
Measure: Number; unit: percentage of participants
Arm/Group | Investigational
Number analyzed (Participants) | 8
percentage of participants | 100

2. Primary Outcome: Procedural Technical Success
Description: Successful robotic delivery and retraction of all PCI devices during CorPath PCI procedure.
Time Frame: Intervention
Population: Total number of PCI devices.
Measure: Number; unit: percentage of PCI devices
Arm/Group | Investigational
Number analyzed (Participants) | 8
percentage of PCI devices | 97.8

ADVERSE EVENTS:
Arm/Group | Investigational
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No